CLINICAL TRIAL: NCT03683758
Title: Effects of the FIFA11+ Warm-up Program on Speed, Agility, and Vertical Jump Performance in Adult Female Amateur Soccer Players
Acronym: FIFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: North Shore Girls Soccer Club (Unknown)
Responsible Party: Principal Investigator, Cheryl Beach, Adjunct Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H18-00383
Record Dates: First submitted 2018-09-10; First posted 2018-09-25 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Soccer; Exercise; Athletic Performance
Keywords: football; soccer; warm-up; FIFA; 11+; performance; speed; agility; jump
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A parallel, two-group, pre-post comparative trial is proposed for this study. Two soccer teams comprise the convenience sample. One team ("Impact") will be allocated to the control group while the other team ("Hearts") are allocated to the intervention group. Participant allocation is premeditated due to Dr. Matt Wentzell's regular paramedical involvement with the "Hearts" and therefore his ability to oversee and administer the intervention warm-up. The control warm-up will be run by the coaching staff of the control group.
  Performance pre-testing will be performed by three trained assistants one week after the 2018/2019 soccer season begins. Tests will be performed three times with the best test score being recorded.
  Both groups will then complete their assigned warm-up three times per week for eight weeks. Both groups will complete posttesting within three days of the trial period concluding in a fashion identical to that of the pre-testing session.
Who Masked: Outcomes Assessor
Masking Description: Participants from both teams will be aware of whether or not they received the intervention warm-up since the intervention warm-up would be a deviation from what each team typically performs for a warm-up.
  Investigator, Dr. Matt Wentzell is not blinded to which group is receiving the intervention warm-up since he will be leading the warm-up over the 8-week period.
  The three trained assistants will be performing the performance pre- and posttesting. They will be blinded to the group each player has been allocated to.
  Any study member that is not blinded will not be performing the pre- and posttesting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA11+ / Intervention Group (Experimental): This group will complete the FIFA11+ warm-up three times per week for eight weeks.
  Interventions: Other: FIFA11+
- Typical Warm-up / Control Group (Active Comparator): This group will complete their usual warm-up three times per week for eight weeks
  Interventions: Other: 'Usual' Soccer Warm-up

INTERVENTIONS:
Other: FIFA11+ — The FIFA11+ has three parts and consist of 15 exercises.
  Part 1 consists of active stretching, running and controlled partner contact drills.
  Part 2 has three difficulty levels for 6 sets of exercises. The exercises consist of core and leg strength exercises, balance and plyometric drills. The exercises in this section are perhaps the most unique element to the FIFA11+ warm-up, as strength-specific exercises like the Nordic Hamstring Curl are not generally included in soccer warm-ups.
  Part 3 consists of higher intensity running drills, compared to those covered in Part 1.
  Unlike many soccer warm-ups, the FIFA11+ has been studied rigorously in terms of its injury reduction potential.
  Arms: FIFA11+ / Intervention Group
Other: 'Usual' Soccer Warm-up — This warm-up is time-matched to the FIFA11+ (approximately 20 minutes) and is considered 'usual' for the team.
  This warm-up consists of stretching, running and agility drills, in addition to "small sided" games with a soccer ball, which is not a part of the FIFA11+.
  The 'usual' warm-up is decided by the coach with no standardization nor any formal research on its effectiveness in injury reduction or performance enhancement.
  Arms: Typical Warm-up / Control Group

SUMMARY:
This study is being conducted for a master's dissertation. Our goal is to determine if there are physical performance benefits to performing the FIFA11+ soccer warm-up program in adult female soccer players over an eight week period. This topic has been studied primarily using male soccer players. The performance effects in adult female soccer players is currently unknown.

This warm-up has been shown to reduce non-contact injury rates in soccer players aged >13. If performance benefits are demonstrated in this study, in addition to the reported injury reduction benefits of the FIFA11+ warm-up, program adherence and player performance could improve.

ELIGIBILITY:
Inclusion Criteria:

* Must be a female amateur soccer players on a North Shore Girls Soccer Club Selects A Team
* Must be between the ages of 18 and 45
* Must play a forward, midfield or defender position

Exclusion Criteria:

* Mustn't play a goal keeper position. The physical demands of this position is drastically different than all other soccer positions. The training effects from practices and games are unique and may therefore influence the effects the FIFA11+ has on players of this particular positions.
* Mustn't have an illness or injury preventing them from participating in soccer practice, games, and testing procedures. Injury or illness would likely result in poorer physical performance outcomes relative to healthy participants.
* Mustn't miss a physical performance testing session. Pre- and posttest data is required to determine if there are changes in performance metrics in relation to both the intervention and control groups.
* Mustn't be pregnant or of childbearing potential for the duration of the study (10 weeks). The PI and Co-Investigators are not familiar with each participant's reproductive health and history or how pregnancy may affect each participant's response to either the intervention or control group. It is therefore decided that participants that are pregnant or of childbearing potential will be removed from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew N Wentzell, DC, Study Director — University of British Columbia Masters Student; Cheryl Beach, PhD, Principal Investigator — University of British Columbia Faculty of Medicine
Locations (1):
- Windsor Bubble, North Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daneshjoo A, Mokhtar AH, Rahnama N, Yusof A. Effects of the 11+ and Harmoknee Warm-up Programs on Physical Performance Measures in Professional Soccer Players. J Sports Sci Med. 2013 Sep 1;12(3):489-96. eCollection 2013. PMID 24149156
- [Background] Impellizzeri FM, Bizzini M, Dvorak J, Pellegrini B, Schena F, Junge A. Physiological and performance responses to the FIFA 11+ (part 2): a randomised controlled trial on the training effects. J Sports Sci. 2013;31(13):1491-502. doi: 10.1080/02640414.2013.802926. Epub 2013 Jul 16. PMID 23855764
- [Background] Ayala F, Pomares-Noguera C, Robles-Palazon FJ, Del Pilar Garcia-Vaquero M, Ruiz-Perez I, Hernandez-Sanchez S, De Ste Croix M. Training Effects of the FIFA 11+ and Harmoknee on Several Neuromuscular Parameters of Physical Performance Measures. Int J Sports Med. 2017 Apr;38(4):278-289. doi: 10.1055/s-0042-121260. Epub 2017 Feb 13. PMID 28192831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed through convenience sampling. Potential study participants are identified through Co-Investigator, Dr. Matt Wentzell's, prior involvement as the trainer/first aid respondent for one of the two NSGSC teams.
Pre-assignment Details: Participants allocation is premeditated by team-based on the MW's regular paramedical involvement with one of the teams and therefore his ability to oversee and administer the intervention warm-up.
  Goaltenders, pregnancy, injury/illness preventing participation in performance testing, practices or games are all grounds for study exclusion.
Groups:
- FIFA11+ / Intervention Group: This group will complete the FIFA11+ warm-up three times per week for eight weeks.
  FIFA11+: The FIFA11+ has three parts and consist of 15 exercises.
  Part 1 consists of active stretching, running and controlled partner contact drills.
  Part 2 has three difficulty levels for 6 sets of exercises. The exercises consist of core and leg strength exercises, balance and plyometric drills. The exercises in this section are perhaps the most unique element to the FIFA11+ warm-up, as strength-specific exercises like the Nordic Hamstring Curl are not generally included in soccer warm-ups.
  Part 3 consists of higher intensity running drills, compared to those covered in Part 1.
  Unlike many soccer warm-ups, the FIFA11+ has been studied rigorously in terms of its injury reduction potential.
- Typical Warm-up / Control Group: This group will complete their usual warm-up three times per week for eight weeks
  'Usual' Soccer Warm-up: This warm-up is time-matched to the FIFA11+ (approximately 20 minutes) and is considered 'usual' for the team.
  This warm-up consists of stretching, running and agility drills, in addition to "small sided" games with a soccer ball, which is not included in the FIFA11+.
  The 'usual' warm-up is decided by the coach with no standardization nor any formal research on its effectiveness in injury reduction or performance enhancement.
Period: Overall Study
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group
Started | 11 | 10
Completed | 8 | 7
Not Completed | 3 | 3
Not completed — Non-study commitment conflict | 1 | 3
Not completed — Illness preventing participation | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Typical Warm-up / Control Group: This group will complete their usual warm-up three times per week for eight weeks
  'Usual' Soccer Warm-up: This warm-up is time-matched to the FIFA11+ (approximately 20 minutes) and is considered 'usual' for the team.
  This warm-up consists of stretching, running and agility drills, in addition to "small sided" games with a soccer ball, which is not a part of the FIFA11+.
  The 'usual' warm-up is decided by the coach with no standardization nor any formal research on its effectiveness in injury reduction or performance enhancement.
- Total: Total of all reporting groups
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (6.6) | 27.1 (3.2) | 27.6 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 10 | 21
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 169.3 (5.4) | 163.3 (5.6) | 166.4 (6.2)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 62.7 (5.7) | 60.2 (8.2) | 61.5 (7.0)
Years of experience [Mean (Standard Deviation); unit: years] | 20.9 (6.3) | 20.1 (1.8) | 20.5 (4.6)
Moderate/high intensity activity per week (hours) [Mean (Standard Deviation); unit: hours] | 7 (3.4) | 6.9 (3.5) | 7.0 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in 10m Sprint Times After an 8 Week Intervention
Description: 10m sprint times will be recorded in seconds.
  The 10m sprint involves a stationary participant starting behind a timing gate and running through a second timing gate 10 meters away.
  Three trials will be performed during the pre-test and the posttest, with the best time being selected for each. Participants will have a 2-minute break between trials.
Time Frame: Intervention is 8 weeks in duration with baseline and post-test outcome measurements occurring within 3 days of the commencement and end of the intervention period
Population: Three players from each team were not included in the analysis due to breach of inclusion criteria (i.e. injury, illness and/or missing a testing session)
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group
Number analyzed (Participants) | 8 | 7
Percentage of change | 4.13 (5.85) | -1.08 (4.38)

2. Primary Outcome: Percentage Change From Baseline in Agility T-Test Times After an 8 Week Intervention
Description: Agility T-test times will be recorded in seconds..
  The Agility T-Test involves a stationary participant running forward through a timing gate to touch a cone 10 yards away, shuffle 5 yards to the left to touch a second cone, shuffle right 10 yards to touch a third cone, shuffle left to touch a fourth cone (the first cone touched after the 10 yard run), then back-peddle 10 yards to pass through the timing gate a second time. This running pattern creates a "T" shape with the vertical and horizontal components of the "T" measuring 10 yards each.
  Three trials will be performed during the pre-test and the posttest, with the best time being selected for each. Participants will have a 2-minute break between trials.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group
Number analyzed (Participants) | 8 | 7
Percentage of change | 8.18 (2.35) | 5.89 (2.12)

3. Primary Outcome: Percentage Change From Baseline in Squat Jump Height After an 8 Week Intervention
Description: Squat jumps will be measured in centimeters.
  This test requires each participant to stand on a contact mat with their hands on their hips, squat and pause in a position with their knees at a 90 degree angle, then propel upward as high as possible.
  Three trials will be performed during the pre-test and the posttest, with the best time being selected for each. Participants will have a 1-minute break between trials.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group
Number analyzed (Participants) | 8 | 7
Percentage of change | 11.88 (6.9) | 7.54 (7.1)

4. Secondary Outcome: Warm-up Attendance
Description: Practice and game attendance will be recorded so warm-up compliance may be calculated. This will be done three days per week for eight weeks.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of warm-ups attended
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group
Number analyzed (Participants) | 8 | 7
Percentage of warm-ups attended | 79.41 (0.09) | 80.36 (0.16)

5. Other Pre Specified Outcome: Player Information
Description: Month and year of birth, height, weight and player position, number of years playing soccer, injury status, approximate number of hours of moderate/high intensity exercise per week (including soccer), and pregnancy status will be collected from each player.
  This information will be collected to compare and contrast the averages of these variables once participants are assigned to the control or intervention group.
Time Frame: 5 minutes before pre-testing.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the pre-testing phase, through the 8 week intervention, up until the end of the post-testing phase for a total of 9 weeks (i.e. up to 3 days before and 3 days after the intervention period).
Description: Adverse event collection was performed for the intervention group via Co-Investigator's (MW) presence at all performance testing sessions and all practices and games over the eight week intervention period.
  Adverse events collection for the control group was performed by monitoring participant attendance on a weekly basis. If three or more warm-ups were missed, Co-Investigator (MW) would follow up with the control group regarding the reason a player may not be in attendance.
Arm/Group | FIFA11+ / Intervention Group | Typical Warm-up / Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIFA11+ / Intervention Group (N=11) | Typical Warm-up / Control Group (N=10)
ACL Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — An ACL tear was sustained by a participant in the FIFA11+ group. The ACL tear did not occur during the intervention warm-up. The participant sustained the injury during a game after returning from a 2-week vacation, voiding her study participation.

LIMITATIONS AND CAVEATS:
This pilot study was under-powered. Time and resources allowed for only two testing sessions which limited participant availability. With additional testing sessions, more players likely could attend participated in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT03683758/Prot_SAP_000.pdf